CLINICAL TRIAL: NCT05506917
Title: Impact of Periodontal Treatment on Brain Hemodynamics
Brief Title: Perio Treatment & Cerebrovascular Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Yago Leira Feijoo, Postoctoral resseacher and clinical supervisor, University of Santiago de Compostela
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT-01
Record Dates: First submitted 2022-08-12; First posted 2022-08-18 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Periodontal Index

STUDY DESIGN:
Intervention Model Description: pre-post comparison study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Periodontal treatment group (Experimental): Patients will receive an intensive (non surgical) regimen of scaling and root planing of the root surfaces under local analgesia (depending on the severity in one session or two sessions within 2 days). Any tooth that from the baseline examination is defined as hopeless or irrational to treat will be extracted at the oral hygiene visit. After the 2 months re-assessment individuals if presenting with at least one periodontal pocket of 6 mm in depth will undergo additional corrective periodontal therapy consisting of periodontal surgery and re-instrumentation under local analgesia. If surgical periodontal therapy is not indicated, appropriate re-instrumentation of the sites will be performed.
  Interventions: Procedure: periodontal treatment

INTERVENTIONS:
Procedure: periodontal treatment — Patients will receive an intensive (non surgical) regimen of scaling and root planing of the root surfaces under local analgesia (depending on the severity in one session or two sessions within 2 days). Any tooth that from the baseline examination is defined as hopeless or irrational to treat will be extracted at the oral hygiene visit. After the 2 months re-assessment individuals if presenting with at least one periodontal pocket of 6 mm in depth will undergo additional corrective periodontal therapy consisting of periodontal surgery and re-instrumentation under local analgesia. If surgical periodontal therapy is not indicated, appropriate re-instrumentation of the sites will be performed.

SUMMARY:
Periodontitis has been linked to increased risk of cerebrovascular disease. Impaired brain hemodynamics has been suggested as early markers of cerebral macro and microangiopathy. Therefore, the aim of this clinical trial will be to assess the potential effect of periodontal treatment on cerebral hemodynamics in otherwise healthy patients with severe periodontitis over 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy subjects with severe periodontitis.

Exclusion Criteria:

* <10 teeth
* current smokers
* undergo periodontal treatment within the last 6 months.
* receive antibiotics or anti-inflammatory drugs within the last 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Cerebrovascular reactivity (CvR) (%) | Baseline-6 months
  CvR to hypercapnia was evaluated by means of the breath-holding index (BHI). Two dual 2-MHz transducers fitted on a headband and placed on the temporal bone windows were used to obtain a bilateral continuous measurement of mean flow velocity in the middle cerebral arteries. Depth of insonation ranged from 48 to 52 mm. The BHI is obtained by dividing the percentage increase in mean flow velocity occurring during breath holding by the length of time (seconds) subjects hold their breath af- ter a normal inspiration ([mean flow velocity at the end of breath holding minus mean flow velocity at rest divided by mean flow velocity at rest] multipled by 100 divided by seconds of breath holding).

SECONDARY OUTCOMES:
Pulsatility index | Baseline-6 months
  Gosling's pulsatility index (PI) of the middle cerebral artery will be calculated according to the following formula: PI = (Vmax -Vmin)/Vmean
Resistivity index | Baseline-6 months
  Resistivity index (RI) of the middle cerebral artery will be calculated according to the following formula: RI = (Vmax -Vmin)/Vmax
Serum high sensitivity C-reactive protein (hs-CRP) | Baseline-6 months
  Levels of hs-CRP in serum will be measured by ELISA (mg/L)
Brachial flow-mediated dilatation | Baseline-6 months
  After detection of brachial artery vasomotion, ultrasound evaluation will be made on the dominant forearm. Two- dimensional brachial artery imaging and measurements were performed in all patients by the same operator. Straight segments of the artery will be chosen above the antecubital fosse, perpendicular to the ultrasound beam and along its long axis. Flow-mediated dilatation caused by shear-induced endothelial nitric oxide production will be detected after occlusion of the forearm circulation. A longitudinal image will be used to measure brachial artery diameter; a blood pressure cuff will be inflated on the upper arm to 300 mmHg for 4 min and then deflated, and after 45 s to 1 min, a second longitudinal scan will be obtained, to calculate the brachial artery diameter.
Carotid intima-media thickness | Baseline-6 months
  The image will be focused on the posterior (far) wall of the left carotid artery. A minimum of four measurements of the common carotid far wall was taken 10 mm proximal to the bifurcation, to derive the mean carotid intima-media thickness. The presence of an atheroma plaque will be evaluated in the common and internal carotid extracranial arteries as well as the bifurcations according to standardized scanning and reading protocols. Plaque will be defined as a focal structure that encroaches into the arterial lumen at least 0.5 mm or 50% of the surrounding intima-media thickness value, or demonstrates a thickness >1.5 mm as measured from the media-adventitia interface to the intima- lumen interface.
Probing pocket depth | Baseline-3 months-6 months
  Will be measured from the free gingival margin to the bottom of the sulcus or pocket (in mm)
Clinical attachment level | Baseline-3 months-6 months
  measured from the cemento-enamel junction (CEJ) to the bottom of the sulcus or pocket (in mm)
Full-mouth bleeding score | Baseline-3 months-6 months
  Defined as the number of sites with gingival bleeding on probing (BoP) divided by the total number of sites per mouth, multiplied by 100 (%)
Full-mouth plaque score | Baseline-3 months-6 months
  Defined as the number of sites with detectable supragingival dental plaque divided by the total number of sites per mouth, multiplied by 100 (%)

CONTACTS AND LOCATIONS:
Overall Officials: Yago Leira, PhD, Principal Investigator — University of Santiago de Compostela
Locations (1):
- University of Santiago de Compostela, Santiago de Compostela, Spain

IPD SHARING:
Plan to Share IPD: No
only upon request to PI